CLINICAL TRIAL: NCT04985968
Title: A Randomised Double-Blind Placebo-Controlled Phase III Clinical Study to Evaluate the Efficacy and Safety of Cobitolimod as an Induction and Maintenance Therapy in Participants With Moderate to Severe Active Left-Sided Ulcerative Colitis
Brief Title: The Efficacy and Safety of Cobitolimod in Participants With Moderate to Severe Active Left-Sided Ulcerative Colitis
Acronym: CONCLUDE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to futility
Sponsor: InDex Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSUC-01/21
Record Dates: First submitted 2021-07-22; First posted 2021-08-02 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Ulcerative Colitis
Keywords: Colitis, Ulcerative; Gastrointestinal Disease; Inflammatory Bowel Diseases; Glucocorticosteroids; Anti-Inflammatory Agents; Therapeutic uses; Cobitolimod; Toll like receptor 9 agonist; TLR9 agonist; Kappaproct; IDX0150; DIMS0150
MeSH Terms: conditions — Colitis, Ulcerative; Gastrointestinal Diseases; Inflammatory Bowel Diseases | interventions — cobitolimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cobitolimod 250 mg (Experimental): Dose of 250 mg cobitolimod
  2 treatments during induction study and subsequently every third week
  Interventions: Drug: Cobitolimod 250 mg
- Cobitolimod 500 mg (Experimental): Dose of 500 mg cobitolimod
  2 treatments during induction study and subsequently every third week
  Interventions: Drug: Cobitolimod 500 mg
- Placebo (Placebo Comparator): Dose of Placebo
  2 treatments during induction study and subsequently every third week
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cobitolimod 250 mg — Rectal administration
  Other Names: Kappaproct
  Arms: Cobitolimod 250 mg
Drug: Cobitolimod 500 mg — Rectal administration
  Other Names: Kappaproct
  Arms: Cobitolimod 500 mg
Drug: Placebo — Rectal administration
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the efficacy of cobitolimod treatment compared to placebo in inducing clinical remission, in participants with moderate to severe active left-sided UC and to evaluate the efficacy of cobitolimod maintenance treatment compared to placebo in inducing or maintaining clinical remission at week 52, in participants with clinical response at week 6 after induction treatment with cobitolimod.

DETAILED DESCRIPTION:
This phase III study protocol includes an induction study for 6 weeks and a maintenance study for an additional 45 weeks.

In the induction study there will be an initial phase to explore the best dose, between cobitolimod 250 mg and cobitolimod 500 mg using adaptive design.

ELIGIBILITY:
Inclusion Criteria Induction:

* Male or female ≥ 18 years of age.
* Established diagnosis of UC.
* Moderate to severe active left-sided UC assessed by central reading.
* Have inadequate response, loss of response or be intolerant of at least one of the following treatments: Oral GCS, AZA/6-MP, Biologics, JAK-inhibitors, or other approved advanced therapies for UC.
* Allowed to receive a therapeutic dose of the following UC drugs during the study: Oral GCS therapy (≤20 mg prednisone or equivalent/day) , Oral 5-ASA/SP compounds, AZA/6-MP.
* Ability to understand the treatment, willingness to comply with all study requirements, and ability to provide informed consent.

Exclusion Criteria Induction:

* Suspicion of differential diagnosis.
* Acute fulminant UC and/or signs of systemic toxicity.
* UC limited to the rectum or extending beyond the splenic flexure.
* Have failed treatment with more than three advanced therapies of two different therapeutic classes.
* Have had surgery for treatment of UC.
* History of malignancy, unless treated with no relapse of the disease and ≥ 5 years since last treatment (cured).
* History or presence of any clinically significant disorder.
* Concomitant treatment with cyclosporine, methotrexate, tacrolimus, or advanced therapies or similar immunosuppressants and immunomodulators.
* Treatment with rectal GCS, 5-ASA/SP or tacrolimus.
* Long-term treatment (>14 days) with antibiotics or NSAIDs .
* Serious known active infection including history of latent or active tuberculosis.
* Gastrointestinal infections including positive Clostridium difficile stool assay.
* Females who are lactating or have a positive serum pregnancy test.
* Women of childbearing potential not using highly effective contraceptive methods.
* Concurrent participation in another clinical study.
* Previous exposure to cobitolimod.

Inclusion Criteria Maintenance:

* Participants are eligible to be included in the maintenance study if they have achieved clinical response at week 6 and have adhered to the protocol procedures of the induction study.

Exclusion Criteria Maintenance:

* Participants will not be eligible for the maintenance study if they are not willing to comply with all further study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2021-11-24 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Induction - Proportion of participants with clinical remission. | Week 6
  Clinical remission defined by the 3-component Mayo score.
Maintenance - Proportion of participants with clinical remission. | Week 52
  Clinical remission defined by the 3-component Mayo score.

SECONDARY OUTCOMES:
Induction - Proportion of participants with endoscopic improvement. | Week 6
  Endoscopic improvement defined by the Mayo Endoscopic score.
Induction - Proportion of participants with symptomatic remission. | Week 6
  Symptomatic remission defined by the 2-component Mayo score.
Induction - Proportion of participants with clinical response. | Week 6
  Clinical remission defined by the 3-component Mayo score.
Induction - Proportion of participants with normalisation of stool frequency. | Week 6
  Stool frequency defined by the Mayo score for Stool Frequency.
Induction - Proportion of participants with absence of rectal bleeding. | Week 6
  Rectal bleeding defined by the Mayo score for Rectal Bleeding.
Induction - Mean stool frequency. | Week 6
  Mean stool frequency defined by the Mayo score for Stool Frequency.
Induction - Proportion of participants with histologic improvement. | Week 6
  Defined by the Robarts Histologic Index.
Induction - Proportion of participants with histologic remission. | Week 6
  Histologic remission defined by the Robarts Histologic Index.
Induction - Proportion of participants with mucosal healing. | Week 6
  Mucosal healing defined by the Mayo Endoscopic score and Robarts Histologic Index.
Induction - Mean ln-transformed faecal calprotectin. | Week 6
  Mean ln-transformed faecal calprotectin defined by faecal calprotectin values.
Induction - Mean 3-component and 4-component Mayo scores. | Week 6
  Defined by 3-component and 4-component Mayo scores.
Induction - Mean IBDQ total score. | Week 6
  Defined by the Inflammatory Bowel Disease Questionnaire (IBDQ).
Induction - Proportion of participants with an improvement in IBDQ total score. | Week 6
  Defined by the IBDQ.
Maintenance - Proportion of participants with endoscopic improvement. | Week 52
  Endoscopic improvement defined by the Mayo Endoscopic score.
Maintenance - Proportion of participants with clinical remission and steroid-free. | Week 52
  Defined by the 3-component Mayo score and use of glucocorticosteroids.
Maintenance - Proportion of participants with clinical remission among those who achieved clinical remission | Week 52
  Defined by the 3-component Mayo score.
Maintenance - Proportion of participants with symptomatic remission. | Week 52
  Symptomatic remission defined by the 2-component Mayo score.
Maintenance - Proportion of participants with histologic improvement. | Week 52
  Histologic improvement defined by the Robarts Histologic Index.
Maintenance - Proportion of participants with histologic remission. | Week 52
  Histologic remission defined by the Robarts Histologic Index.
Maintenance - Proportion of participants with mucosal healing. | Week 52
  Mucosal healing defined by the Mayo Endoscopic score and Robarts Histologic Index.
Maintenance - Proportion of participants with clinical response. | Week 52
  Clinical response defined by the 3-component Mayo score.
Maintenance - Proportion of participants with absence of rectal bleeding. | Week 52
  Rectal bleeding defined by the Mayo score for Rectal Bleeding.
Maintenance - Proportion of participants with normalisation of stool frequency. | Week 52
  Stool frequency defined by the Mayo score for Stool Frequency.
Maintenance - Mean stool frequency. | Week 52
  Mean stool frequency defined by the Mayo score for Stool Frequency.
Maintenance - Mean ln-transformed faecal calprotectin. | Week 52
  Mean ln-transformed faecal calprotectin.
Maintenance - Mean 3-component and 4-component Mayo scores. | Week 52
  Defined by 3-component and 4-component Mayo scores.
Maintenance - Mean IBDQ total score. | Week 52
  Defined by the use of the Inflammatory Bowel Disease Questionnaire (IBDQ).
Maintenance - Proportion of participants with an improvement in IBDQ total score. | Week 52
  Defined by the IBDQ.

CONTACTS AND LOCATIONS:
Overall Officials: Raja Atreya, Professor, Principal Investigator — Friedrich-Alexander University Erlangen-Nuremberg
Locations (203):
- United States (25):
  - Amicis Research Center, Granada Hills, California
  - Allameh Medical Corporation, Mission Viejo, California
  - Prospective Research Innovations Inc., Rancho Cucamonga, California
  - Valiance Clinical Research, Tarzana, California
  - RecioMed Clinical Research Network, Inc., Boynton Beach, Florida
  - MB & V Medical Research, Doral, Florida
  - A+ Research, Inc., Miami, Florida
  - SouthCoast Research Center, Inc, Miami, Florida
  - I.V.A.M. Clinical & Investigational Center LLC, Miami, Florida
  - D&H National Research Centers, Inc., Miami, Florida
  - Medical Professionals Clinical Research Center, Miami, Florida
  - Gastroenterology Group Of Naples, Naples, Florida
  - Alliance Clinical Research - Gastroenterology, Tampa, Florida
  - Cotton O'Neil Clinical Research Center, Topeka, Kansas
  - Clinical Research Institute of Michigan, Troy, Michigan
  - Lenox Hill Hospital, New York, New York
  - Carolina Digestive Health Associates, PA, Charlotte, North Carolina
  - Carolina Research, Greenville, North Carolina
  - Peters Medical Research, High Point, North Carolina
  - Dayton Gastroenterology, Beavercreek, Ohio
  - Digestive Health Associates of Texas, PA, Carrollton, Texas
  - Clinical Research Solution: Digestive Health Associates, Houston, Texas
  - Baylor College of Medicine - Gastroeneterology, Houston, Texas
  - Gastroenterology Associates of Northern Virginia, Fairfax, Virginia
  - Wisconsin Center For Advanced Research, Milwaukee, Wisconsin
- Australia (6):
  - Monash Health, Clayton
  - St Vincent's Hospital Melbourne, Fitzroy
  - The Alfred Hospital, Melbourne
  - Royal Melbourne Hospital, Parkville
  - Mater Health Services, South Brisbane
  - Princess Alexandra Hospital, Woolloongabba
- Austria (4):
  - MedUn Innsbruck, Innsbruck
  - LKH Klagenfurt, Klagenfurt
  - Universitätsklinikum Salzburg, Salzburg
  - Akh Wien, Vienna
- Belgium (6):
  - UZ Antwerpen, Antwerp
  - Imelda Ziekenhuis, Bonheiden
  - Erasme University Hospital, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - AZ Groeninge - Campus Kennedylaan, Kortrijk
  - AZ Delta, Roeselare
- Bosnia and Herzegovina (8):
  - University Clinical Centre of the Republic of Srpska - Gastroenterology, Banja Luka
  - The University Hospital Foca, Foča
  - Clinical Center University of Sarajevo - Gastroenterology, Sarajevo
  - General Hospital "Prim.dr.Abdulah Nakas", Sarajevo
  - Polyclinic Dr. Al-Tawil, Sarajevo
  - Opca Bolnica Tesanj, Tešanj
  - Plava Medical Group, Tuzla
  - Cantonal Hospital Zenica, Zenica
- Brazil (6):
  - Instituto Goiano de Gastroenterologia e Endoscopia Digestiva Ltda, Goiânia
  - Hospital de Clinicas de Porto Alegre - Centro de Pesquisa Clinica, Porto Alegre
  - Ufrj - Hospital Universitario Clementino Fraga Filho, Rio de Janeiro
  - Praxis Pesquisa Medica, Santo André
  - CEMEC - Centro Multidisciplinar de Estudos Clinicos, São Bernardo do Campo
  - Kaiser Clinica, São José do Rio Preto
- Canada (3):
  - MUMC - Hamilton Health Sciences, Hamilton
  - Installation Hospital Maisonneuve-Rosemont, Montreal
  - Royal University Hospital, Saskatoon
- Croatia (6):
  - Opca bolnica Bjelovar, Bjelovar
  - Clinical Hospital Osijek, Osijek
  - Opca bolnica Pula, Pula
  - Zadar General Hospital, Zadar
  - Poliklinika Solmed, Zagreb
  - University Hospital Centre Zagreb, Zagreb
- Denmark (5):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Herlev Hospital, Herlev
  - Hillerod Hospital, Hillerød
  - Lillebælt Hospital Vejle, Vejle
- France (11):
  - CHRU de Lille - Hôpital Claude Huriez, Lille
  - CHRU Montpellier-Hopital Saint Eloi - Hepato-gastro-enterologie, Montpellier
  - CHU de Nancy Brabois, Nancy
  - CHU de Nice - Hôpital de l'Archet II - Gastro-Entérologie, Hépatologie, Nice
  - Hopital Bichat - Gastroenterology, Paris
  - Hopital Saint Antoine, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - CHU de Saint Etienne, Hôpital Nord - Service de Gastroentérologie, Saint-Etienne
  - CHU Amiens - Hopital Sud - Service Hepato-Gastroenterolog, Salouël
  - Centre Hospitalier Universitaire de Toulouse - Hopital Rangueil, Toulouse
- Georgia (2):
  - JSC " Evex Hospitals", Batumi
  - LTD Israel-Georgian Medical Research Clinic Helsicore, Tbilisi
- Germany (16):
  - Universitätsklinikum Augsburg, Augsburg
  - Charité - Universitätsmedizin Berlin KöR, Berlin
  - University Hospital Cologne AöR, Cologne
  - MVZ Sanaklinikum Duisburg, Duisburg
  - Universitätsklinikum Erlangen, Erlangen
  - Agaplesion Markus Krankenhaus, Frankfurt am Main
  - Klinikum der Johann Wolfgang Goethe-Universität - Medizinische Klinik I, Frankfurt am Main
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Uniklinik Halle (Saale), Halle
  - Gastroenterology Outpatient Clinic Prof. Dr. med. Ehehalt, Heidelberg
  - University Hospital Schleswig-Holstein, Kiel
  - Universitätsmedizin Mannheim, Mannheim
  - Medius Klinik Nürtingen, Nürtingen
  - Universitätsklinikum Rostock, Rostock
  - Universitätsklinikum Ulm, Ulm
  - Internistische Praxis Weyhe, Weyhe
- Hungary (5):
  - Clinexpert Egészségügyi Szolgáltató És Kereskedelmi Kft., Budapest
  - Pannónia Magánorvosi Centrum Kft, Budapest
  - Semmelweis Egyetem Altalanos Orvostudomanyi Kar Sebeszeti, Transzplantacios es Gasztroenterologiai Klinika, Budapest
  - Semmelweis Egyetem Altalanos Orvostudomanyi Kar, Budapest
  - SzTE Szt-Gy A Orvostud Kar Bel Klin, Szeged
- Israel (6):
  - The Barzilai Medical Center, Ashkelon
  - The Edith Wolfson Medical Center, Holon
  - Hadassah Medical Organization, Hadassah Medical Center, Ein-, Jerusalem
  - Shaare Zedek Medical Center, Jerusalem
  - Galilee Medical Center (Western Galilee Hospital), Nahariya
  - Kaplan Medical Center, Rehovot
- Italy (12):
  - ASST Papa Giovanni XXIII - Cardiologia - Bergamo, Bergamo
  - AO Brotzu, Cagliari
  - Universita degli Studi di Firenze - Azienda Ospedaliero - Un, Florence
  - IRCCS Ospedale San Raffaele, Milan
  - Azienda Ospedaliera San Gerardo, Monza
  - AOU di Padova, Padua
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata (P, Roma
  - Policlinico Universitario Agostino Gemelli, Roma
  - Policlinico Universitario Campus Biomedico, Rome
  - A.O. Ordine Mauriziano Di Torino, Torino
  - AOU S. Maria della Misericordia, Udine
  - Universita degli Studi dell'Insubria - Ospedale di Circolo e, Varese
- Lithuania (5):
  - Hospital of Lithuanian University of Health Sciences Kauno Klinikos, Kaunas
  - Klaipeda Seamen's Hospital, Klaipėda
  - Republic Klaipeda Hospital, Klaipėda
  - Panevezio ligonine, Panevezys
  - Vilniaus Universiteto ligonines Santariskiu Klinikos, Vilnius
- Mexico (5):
  - Instituto de Investigaciones Aplicadas a la Neurociencia A.C., Durango
  - Clinicos Asociados Bocm, S.C., Mexico City
  - Medical Care and Research S. A. de C. V, Mérida
  - Centro Regiomontano de Estudios Clinicos Roma SC, Monterrey
  - Clinical Research Institute S.C., Tlalnepantla
- Radboud University Medical Center, Nijmegen, Netherlands
- Norway (4):
  - Ålesund Hospital, Møre & Romsdal Hospital trust, Dept. of Medicine, div of Gastroenterology and the Clinical research unit HMR, Ålesund
  - Akershus Universitetssykehus, Lørenskog
  - Universitetssykehuset Nord-Norge Tromsø, Gastrolab, Medisinsk poliklinikk, B8, Tromsø
  - Vestfold Hjertesenter As, Tønsberg
- Poland (19):
  - MPS - MED sp. z o.o., Grudziądz
  - MZ Badania Slowik Zymla Spolka jawna, Knurów
  - Centrum Medyczne Plejady, Krakow
  - Centrum Medyczne PROMED, Krakow
  - Krakowskie Centrum Medyczne Sp. z o.o., Krakow
  - Szpital Zakonu Bonifratrow Sw. Jana Bozego w Lodzi, Lodz
  - Klinika Badawcza Centrum Badawcze Panaceum Agnieszka Brzezicka, Magdalena Lenkiewicz Sp. z o.o., Malbork
  - Twoja Przychodnia - Opolskie Centrum Medyczne, Opole
  - Medicome Sp. z o.o., Oświęcim
  - Szpital Kliniczny im. Heliodora Swiecickiego Uniwersytetu Medycznego im. Karola Marcinkowskiego w Poznaniu, Poznan
  - ETG Skierniewice, Skierniewice
  - KO-MED Centra Kliniczne Staszow, Staszów
  - Twoja Przychodnia - SCM, Szczecin
  - GASTROMED Kopoń, Zmudziński i Wspólnicy spółka jawna, Specjalistyczne Centrum Gastrologii i Endoskopii, Specjalistyczne Gabinety Lekarskie, Torun
  - Bodyclinic sp. z o.o. sp.k., Warsaw
  - Centralny Szpital Kliniczny MSWiA w Warszawie, Warsaw
  - Centrum Zdrowia Matki, Dziecka i Mlodziezy, Warsaw
  - PlanetMed, Wroclaw
  - ETG Zamosc, Zamość
- Portugal (4):
  - Hospital Prof. Doutor Fernando Fonseca (HFF) (Hospital Amadora Sintra), Amadora
  - Hospital de Braga, Braga
  - Hospital Beatriz Angelo (HBA), Loures
  - Centro Hospitalar de Entre o Douro e Vouga (CHEDV)- Hospital São Sebastião, Santa Maria da Feira
- Romania (6):
  - Sana Monitoring, Bucharest
  - Spitalul Clinic Colentina, Bucharest
  - Spitalul Clinic Judetean de Urgenta Cluj-Napoca, Cluj-Napoca
  - Spitalul Clinic Judetean de Urgenta "Sf. Spiridon" Iasi, Iași
  - Spitalul Clinic Judetean Mures, Târgu Mureş
  - Cabinet Particular Policlinic Algomed, Timișoara
- Serbia (7):
  - Clinic Center of Serbia, Belgrade
  - Clinical Hospital Center "Dr. Dragisa Misovic", Belgrade
  - Euromedik Hospital, Belgrade
  - Zvezdara University Medical Center, Belgrade
  - Clinical Center Kragujevac - Center for Gastroenterohepatology, Kragujevac
  - General Hospital Dr Djordje Joanovic, Zrenjanin
  - General hospital Zrenjanin, Zrenjanin
- Slovakia (5):
  - FNsP F.D.R. Banska Bystrica, Banská Bystrica
  - CLINIQ s.r.o., Bratislava
  - ENDOMED s.r.o., Košice
  - GASTROMEDIC, s.r.o., Nové Zámky
  - Accout Center s.r.o., Šahy
- South Korea (10):
  - Inje University Haeundae Paik Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Hanyang University Guri Hospital, Guri-si
  - Kyung Hee University Hospital, Seoul
  - Seoul National University Bundang Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Kyung Hee University Hospital - Internal Medicine, Soeul
  - Kyung Hee University Hospital, Soeul
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon
  - Yonsei University, Wonju Severance Christian Hospital, Wŏnju
- Sweden (3):
  - Örebro Univ. Hospital, Örebro
  - Karolinska Universitetssjukhuset - Gastroenterology, Stockholm
  - Uppsala University Hospital, Akademiska, Uppsala
- Turkey (Türkiye) (3):
  - Hacettepe University Medical Faculty - Hematology, Ankara
  - Istanbul University Medical Faculty, Istanbul
  - Mersin Universtiy Medical Faculty, Mersin
- United Kingdom (10):
  - Northern Care Alliance NHS Foundation Trust-Fairfield General Hospital - Gastroenterology, Bury
  - Accellacare Warwickshire Quality Research Site, Coventry
  - County Durham and Darlington NHS Foundation Trust (CDDFT) - Darlington Memorial Hospital, Darlington
  - Glasgow Royal Infirmary, Glasgow
  - North West London Hospitals NHS Trust, Harrow
  - Central Middlesex Hospital, London
  - Kings College Hospital, London
  - Accellacare North London, Northwood
  - Accellacare Limited/Accellacare of South London, Orpington
  - Royal Berkshire Hospital, Reading

IPD SHARING:
Plan to Share IPD: No